CLINICAL TRIAL: NCT02728648
Title: Population Pharmacokinetic-Pharmacodynamic Study of Intravenous Oxycodone in Malaysian Population
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Malaya (Other)
Responsible Party: Principal Investigator, Chaw Sook Hui, Dr, University of Malaya
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20162-2143
Record Dates: First submitted 2016-03-25; First posted 2016-04-05 (Estimated); Last update posted 2022-01-28 (Actual); Status verified 2022-01

CONDITIONS: Pain
Keywords: Pain Management; Pharmacokinetics; Pharmacodynamics
MeSH Terms: conditions — Pain; Agnosia | interventions — Oxycodone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Active (Other): Open label IV Oxycodone 0.1 mg/kg Bolus Pharmacokinetic-Pharmacodynamic Study
  Interventions: Drug: Oxycodone

INTERVENTIONS:
Drug: Oxycodone — Pain Management
  Other Names: OxyNorm

SUMMARY:
Oxycodone has been in clinical use for decades. It is an effective alternative to morphine for moderate to severe acute or chronic pain and has been found to improve quality of life. The drug has been used parenterally or orally as perioperative analgesia or for cancer pain relief. Despite its long clinical experience, prescribing errors and misuse may lead to addiction and accidental overdose. Currently, little is known about the pharmacokinetic properties of intravenous oxycodone among paediatric patients in this region even though the drug has been used in children in other countries such as Finland. Therefore, a pharmacokinetic-pharmacodynamic study of oxycodone among Malaysian pediatric patients is warranted.

DETAILED DESCRIPTION:
Oxycodone (14-hydroxy-7,8 dihydrocodeinone) is a strong, semisynthetic thebaine derivative µ-opioid receptor agonist. This drug is an effective alternative to morphine for moderate-to-severe pain. Oxycodone has been used parenterally or orally for perioperative analgesia or for cancer pain relief. The drug has a longer analgesic action than morphine. In terms of analgesic potency, intravenous oxycodone is about 1.6 times

The adverse effects of oxycodone are mostly similar to those of other opioids. Oxycodone, however, does not cause histamine release. The drug induces less nausea and vomiting, less sedating, and less central nervous system excitatory effects than morphine.

A large between-subject variability in pharmacokinetic properties of oxycodone has been observed. The variability could be attributed to the different body size and age-related difference in drug elimination organ system function. A 2-compartment first-order open model describes oxycodone pharmacokinetics in Finnish children (age 5.4±2.1 years) after an intravenous bolus dose of 0.1 mg kg-1 for post ophthalmic surgery pain relief. The authors reported a mean clearance (CL) and the steady-state volume of distribution (Vss) of oxycodone 15.2 mL min-1 kg-1 (0.912 L h-1 kg-1) and 2.1 L kg-1 respectively. A greater ventilator depression than comparable analgesic doses of other opioids was also observed. A pharmacokinetic study carried out in 9 young Finnish adult surgical patients reveals a clearance of 0.78 L min-1 (46.8 L h-1) and a volume of distribution (V) of 2.60 L kg-1. The mean area under the curve (AUC)( t=0,12) ratio of noroxycodone (main metabolite) to oxycodone is 0.33. In a study on 69 Japanese adults (mean age 66 years, mean weight 52.8 kg) receiving intravenous oxycodone for cancer pain relief, a one-compartment first-order open model describes the pharmacokinetics of oxycodone. The mean CL and volume of distribution (V) are 24.6 L h-1 and 214 L or 4.053 L kg-1.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 3 to 65 years
* Generally healthy as documented by medical history (ASA 1-II)
* Opioid-naïve
* Patient is scheduled for a surgical procedure/procedures that is/are expected to require an analgesia with an opiate level medication.
* Patient who will remain hospitalized for at least 24 hours after dosing with the study drug.
* A negative urine pregnancy test at screening for females of childbearing potential

Exclusion Criteria:

* Patient is a lactating or breastfeeding female
* Patient has known allergy to oxycodone or any ingredient in oxycodone dosage form.

Ages: 3 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Clearance (CL) | 18 months
  Clearance: volume of plasma from which oxycodone is completely removed per unit time;

SECONDARY OUTCOMES:
Volume of distribution of IV oxycodone | 18 months
  Volume of distribution: theoretical volume that would be necessary to contain the total amount of oxycodone at the same concentration that it is observed in the blood plasma.

CONTACTS AND LOCATIONS:
Overall Officials: Sook Hui Chaw, M.Med, Principal Investigator — University of Malaya
Locations (1):
- Faculty of Medicine, University of Malaya, Kuala Lumpur, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: Yes
Oxycodone pharmacokinetics data
Supporting Information: Study Protocol, SAP
Time Frame: After 5 years of study completion
Access Criteria: Request from primary investigator

REFERENCES:
- [Background] Kalso E, Poyhia R, Onnela P, Linko K, Tigerstedt I, Tammisto T. Intravenous morphine and oxycodone for pain after abdominal surgery. Acta Anaesthesiol Scand. 1991 Oct;35(7):642-6. doi: 10.1111/j.1399-6576.1991.tb03364.x. PMID 1785245
- [Background] Olkkola KT, Hamunen K, Seppala T, Maunuksela EL. Pharmacokinetics and ventilatory effects of intravenous oxycodone in postoperative children. Br J Clin Pharmacol. 1994 Jul;38(1):71-6. doi: 10.1111/j.1365-2125.1994.tb04324.x. PMID 7605420
- [Background] Poyhia R, Olkkola KT, Seppala T, Kalso E. The pharmacokinetics of oxycodone after intravenous injection in adults. Br J Clin Pharmacol. 1991 Oct;32(4):516-8. doi: 10.1111/j.1365-2125.1991.tb03942.x. PMID 1958450
- [Background] Kokubun H, Yoshimoto T, Hojo M, Fukumura K, Matoba M. Pharmacokinetics of oxycodone after intravenous and subcutaneous administration in Japanese patients with cancer pain. J Pain Palliat Care Pharmacother. 2014 Dec;28(4):338-50. doi: 10.3109/15360288.2014.969872. Epub 2014 Oct 31. PMID 25359452